CLINICAL TRIAL: NCT06815159
Title: Tissue Markers Predictive of Early Stenosis in the Arterovenous Fistula for Hemodialysis
Acronym: FAV-2019
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FAV-2019
Record Dates: First submitted 2024-11-28; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-11

CONDITIONS: AV Fistula
MeSH Terms: conditions — Arteriovenous Fistula | interventions — Dialysis

STUDY DESIGN:
Intervention Model Description: The study involves the recruitment of two populations. POPULATION 1 (surgical sample of excess venous segment): at least 75 consecutive patients, enrolled according to the inclusion criteria and subjected to first AVF surgery
  POPULATION 2 (surgical sample of arterialized venous segment from removal of previous AVF): at least 75 consecutive patients, enrolled according to the inclusion criteria and subjected to re-intervention for correction of complication and/or new AVF by proximalization,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- First FAV (Experimental): Group of patient with first FAV
  Interventions: Biological: Identification any tissue markers predictive or favoring early stenosis in AVF for haemodialysis.
- Secondary FAV (Experimental): Group of patients with reintervention of FAV
  Interventions: Biological: Identification any tissue markers predictive or favoring early stenosis in AVF for haemodialysis.

INTERVENTIONS:
Biological: Identification any tissue markers predictive or favoring early stenosis in AVF for haemodialysis. — Primary objective
  1. Identify any predictive or favoring tissue markers of early stenosis in AVF for hemodialysis.
     Secondary objectives
  2. Compare the results on the possible different expression of tissue markers before and during dialysis.
  3. Compare the results on the possible different expression of tissue markers between AVFs made with portions of cephalic vein and AVFs made with portions of basilic vein, in order to evaluate whether the different topographic origin of the AVF can influence its duration.

SUMMARY:
The study involves the recruitment of two populations. POPULATION 1 (surgical sample of excess venous segment): at least 75 consecutive patients, enrolled according to the inclusion criteria and subjected to first AVF surgery as part of the normal care pathway, at the Metropolitan Vascular Surgery Unit, Dir. Prof. Mauro Gargiulo of the S.Orsola-Malpighi University Hospital.

POPULATION 2 (surgical sample of arterialized venous segment from removal of previous AVF): at least 75 consecutive patients, enrolled according to the inclusion criteria and subjected to reoperation for correction of complication and/or new AVF by proximalization, as part of the normal care pathway, at the Metropolitan Vascular Surgery Unit, Dir. Prof. Mauro Gargiulo of the S.Orsola-Malpighi University Hospital.

DETAILED DESCRIPTION:
The following study will enroll two cohorts of patients: 75 patients from Population 1 and 75 patients from Population 2, according to the inclusion criteria. Since this is an exploratory study, this number is considered sufficient to observe and compare tissue markers associated with early AVF stenosis.

Patients will be treated according to clinical practice in accordance with the physician's judgment.

The study includes: the recruitment of patients from the two study populations, the obtaining of the surgical specimen from both populations and its sending to the Pathology Department, as part of the normal care pathway, the execution of three tissue samples at the Pathology Department: (i) a sample frozen in liquid nitrogen and stored in an ultrafreezer at -80°C for RT-PCR analysis; (ii) a sample placed in PBS for cell culture; (iii) the remainder of the sample fixed in formalin, embedded in paraffin and processed according to the normal care pathway and histological diagnosis. 2 µm slices will be cut from the paraffin block for histological staining and histochemical and IIC investigations; execution of cell culture investigations and execution of RT-PCR investigations.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years;
* Patients candidates for first AVF for hemodialysis or correction of AVF complication, as part of the normal care pathway;
* Obtaining informed consent signed by the patient

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-03-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Identify any predictive or favoring tissue markers of early stenosis in AVF for hemodialysis. | From the first patient entrolled, up to the 150th patient, an average of 6 years
  Biomarkers of the treated fistula are histologically examined

SECONDARY OUTCOMES:
Different expression of tissue markers before and during dialysis. | From the first patient enrolled to the 150th patient, an average of 6 years
  Markers expression of the treated tissue are analysed and compared between the two study group.
Markers differences between Basilic and cephalic vein | From the first patient enrolled, up to the 150th patient, up to 6 years
  Compare the results on the possible different expression of tissue markers between AVFs made with portions of cephalic vein and AVFs made with portions of basilic vein, in order to evaluate whether the different topographic origin of the AVF can influence its duration.

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Gargiulo, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS AOU di Bologna Policlinico di Sant'Orsola, Bologna, Italy